CLINICAL TRIAL: NCT07391865
Title: The Effect of Chronotype on Motivation and Academic Achievement in Nursing Students Trained With Flipped Learning Approach: A Randomized Controlled Trial
Brief Title: The Effect of Chronotype on Motivation and Academic Achievement in Students Trained With a Flipped Learning Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Berna Aksoy Kahraman, Assistant Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TÜTF-BAEK 2022/189
Record Dates: First submitted 2025-12-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Nursing students; flipped classroom; traditional training; chronotype; academic performance; motivation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Flipped classroom group (Experimental): The experimental group students were taught the topic titled "Urinary System Applications" based on the flipped classroom approach
  Interventions: Other: Flipped classroom approach
- The traditional classroom approach group (No Intervention): The control group students were taught the topic titled "Urinary System Applications" based on the traditional classroom approach.

INTERVENTIONS:
Other: Flipped classroom approach — The experimental group students were taught the topic titled "Urinary System Applications" based on the FCA. The link to the online education platform required for out-of-class learning in this approach was shared with the students two weeks before the start of the course. Thus, students were able to watch the videos anytime and anywhere at their convenience. The educational platform included 31 videos on urinary system practices, specially prepared by researchers based on Bloom's taxonomy. These videos were organized into 31 sequential and thematically cohesive parts, and each part was interconnected.
  The student could not watch a subsequent part without completing the previous related part. Each video was 10-15 minutes long, with one video introducing the online platform, 27 videos covering the theoretical aspects of the subject, and 3 videos focusing on skill application. Specific questions tailored to the learning outcomes of the subject were embedded in each video. Access to the
  Other Names: Education
  Arms: The Flipped classroom group

SUMMARY:
The rapidly evolving world has influenced the sleep-wake cycles of nursing students, shifting them towards an evening chronotype. This shift has negatively impacted their daytime functionality, motivation, and academic success. Moreover, research indicates that there is an asynchrony between individuals' circadian rhythms and face-to-face classes. Flipped learning can be seen as a potential solution to nursing education. The purpose of this study was to examine the effect of chronotype on motivation and academic achievement in nursing students trained with two different learning approaches.

DETAILED DESCRIPTION:
This study were conducted a randomized controlled experimental design incorporating pre-test and post-test follow-ups. The study sample consisted of volunteer nursing students at the nursing department of a university in western Turkey. In this department, an internship program is offered and the Fundamentals of Nursing course, which is designed to provide 5 hours of theoretical instruction and 8 hours of practical training during the spring semester. The theoretical parts of the courses are conducted in lecture halls using a traditional classroom approach, while the practical parts are carried out in laboratories and clinics. As part of the course, after the instructor delivers the theoretical lecture, students watch videos related to the topic in the lecture hall to enhance their psychomotor skills. The application steps are then explained, followed by hands-on practice in the laboratory.

G*Power 3.1 software was utilized for the power analysis of the study. Based on the study by Aksoy and Gurdoğan, with an effect size of 0.79, a power of 95%, and a significance level of 0.05, it was determined that a minimum of 43 students should be assigned to each group. However, considering a 20% loss rate during the study, it was decided to include at least 52 students in each group. The students were randomly divided into two groups, the experimental and control groups, using the simple randomization method with the Research Randomizer program. A total of 114 students who met the study criteria were assigned to the experimental and control groups, with 57 students in each group. However, three students in the experimental group were excluded from the study because they participated in the training but did not complete the post-training data collection forms. Thus, the study was completed with a total of 111 students, including 57 in the control group and 54 in the experimental group. Turkish version of Morningness-Eveningness Questionnaire and Motivated Strategies for Learning Questionnaire, and theory and skill exams specific to urinary system were used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age,
* To volunteer,
* Taking the Fundamentals of Nursing course for the first time,
* To own a smartphone or computer,
* To have internet access.

Exclusion Criteria:

* Being under 18 years of age,
* Not being a volunteer,
* Having previously taken the Fundamentals of Nursing course,
* Not owning a smartphone or computer.
* Not having internet access.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
The Motivated Strategies for Learning Questionnaire (MSLQ) | Before courses begin and 15 days after the courses concluded, an average of 7 weeks
  The questionnaire was developed by Pintrich et al. in 1991.24 It was adapted to Turkish language by by Büyüköztürk et al. in 2004. This scale allowing students to indicate how well the items describe their personal situation. This scale consists of two main section, learning strategies and motivation, and 15 sub-dimensions. Responses are provided on a 7-point Likert scale, ranging from "not at all true of me" to "very true of me". In this study, the motivation section with its 6 sub-dimensions were applied to the students. Each sub-dimension is scored separately, and increasing scores indicate increased student motivation.
The Morningness-Eveningness Questionnaire (MEQ) | Before courses begin and 15 days after the courses concluded, an average of 7 weeks
  The self-assessment-based form was developed by Horne and Östberg in 1976. The Turkish validity and reliability study was conducted by Pündük et al. in 2005. The form, which is used to determine morningness and eveningness types in the human circadian rhythm, consists of 19 questions. The minimum score that can be obtained from the form is 16, while the maximum score is 86. Based on the total score, individuals are classified as evening type, intermediate type, and morning type. While the Cronbach's alpha value was reported as 0.81 in the study by Pündük et al., it was found to be 0.72 in this study.
The theoretical exam | 15 days after the courses concluded, an average of 7 weeks
  The theoretical exam was developed by the researchers based on the guidelines and standards outlined by the Centers for Disease Control and Prevention. A detailed rubric evaluation was utilized to score student responses. The exam included four open-ended questions. The exam content included questions about the steps of urinary catheterization, types of urinary incontinence and their nursing care, urinary tract infections associated with urinary catheters, and a case study.
The skill exam | 15 days after the courses concluded, an average of 7 weeks
  The skill exam was conducted using a urinary catheterization skill checklist, which consisted of 40 steps and specified the score for each step, prepared based on the literatüre. Both the theoretical and skill exams were graded on a 0-100 scale and were conducted 15 days after the courses concluded. The evaluation were carried out by an independent faculty member who was blinded to the group assignments (experimental or control).

CONTACTS AND LOCATIONS:
Overall Officials: Eylem PASLI GÜRDOĞAN, PhD, Principal Investigator — Trakya University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pintrich, P. R., Smith, D., García, T., McKeachie, W. 1991. A manual for the use of the Motivated Strategies for Learning Questionnaire (MSLQ). University of Michigan.
- [Result] Nam, D., Demircioğlu Diren, D., Horzum, M. B. 2024. Online learning barriers and its relationship to gender, age, work status, and chronotype in university student. Biological Rhythm Research. 55: 260-277. doi: 10.1080/09291016.2024.2336926
- [Result] Büyüköztürk, S., Akgün, Ö. E., Özkahveci, Ö., Demirel, F. 2004. The validity and reliability study of the Turkish version of the motivated strategies for learning questionnaire. Educational Sciences: Theory & Practice. 4: 231-239
- [Result] Balcı, Ö., Çalışkan, M. 2022. Investigation of the relationship between chronotype, learning style and academic achievement of university students during distance education in the pandemic period. Chronobiology International. 39:858-871. doi:10.1080/07420528.2022.2041658
- [Result] Aguilar, R., Santana, M., Larrañeta, B., Cuevas, G. 2021. Flipping the strategic management classroom: Undergraduate students' learning outcomes. Scandinavian Journal of Educational Research. 65:1081-1096. doi:10.1080/00313831.2020.1825524
- [Result] Adan, A., Archer, S. N., Hidalgo, M. P., Di Milia, L., Natale, V., Randler, C. 2012. Circadian typology: a comprehensive review. Chronobiology international. 29:1153-1175. doi:10.3109/07420528.2012.719971